CLINICAL TRIAL: NCT00283257
Title: A Randomized Control Trial That Teaches Oncology Clinical Trial Patients and Their Caregivers Problem Solving Skills.
Brief Title: Simultaneous Care: Linking Palliation to Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 200210794; NCI CA 95260
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Solid Tumor; Lymphoma
Keywords: Problem solving; psychosocial support
MeSH Terms: conditions — Lymphoma

INTERVENTIONS:
Behavioral: Patients and caregivers are taught problem solving skills

SUMMARY:
This is a multi-site randomized control trial taking place at six cancer centers. UC Davis is the lead site. Additional performance sites include the City of Hope Medical Center, Fred Hutchinson Cancer Center at the Univ. of Washington, USC Norris Cancer Center, UCSD Cancer Center, and Johns Hopkins Cancer Center. Clinical trial patients and their caregivers who are randomized to the intervention arm of the study are scheduled for three educational sessions. The sessions focus on teaching problem solving skills based on the COPE problem solving model.

DETAILED DESCRIPTION:
The project introduces and evaluates the effects of a Simultaneous Care Education Intervention, using the COPE model (Creativity, Optimism, Planning and Expert Information) developed by D'Zurilla and Nezu, as one of its key components for cancer patients in Phase I, II and III clinical trials. The SCEI team will use the COPE problem solving educational model to instruct patients on how to problem solve and manage challenges associated not only with the investigational therapy, but also the psychosocial issues that arise from cancer diagnosis, disease progression, treatment, and disease or treatment related symptoms. The educational intervention also sets up a system for regularly contacting the patient and caregiver in order to reinforce what is taught. Patients and caregivers randomized to the intervention arm will receive three education sessions. Patients and designated caregiver will be asked to complete the set of measurement tools approximately every 30 days while enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, must have caregiver who is willing to participate, must be entering a phase 1-3 oncology clinical trial. Must be able to complete first educational session on or before treatment start date. Solid tumor or lymphoma only.

Exclusion Criteria:

* Non-English speaking, no caregiver available, unable to complete first educational session on or before treatment start date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2002-02 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Carducci, M.D., Principal Investigator — Johns Hopkins University; Betty Ferrell, Ph.D, Principal Investigator — City of Hope Medical Center; Anthony Back, M.D., Principal Investigator — Fred Hutchinson Cancer Center, Univ. of Washington; Heinz Josef Lenz, M.D., Principal Investigator — USC Norris Cancer Center; Joanne Mortimer, M.D., Principal Investigator — University of California, San Diego; Frederick J Meyers, MD, Study Chair — University of California, Davis
Locations (1):
- UC Davis Cancer Center, Sacramento, California, United States